CLINICAL TRIAL: NCT04686032
Title: Effect of Early Physical Therapy Interventions on Post-operative Recovery and Complications Following Abdominal Hysterectomy
Brief Title: Effect of Early Rehabilitation on Recovery Following Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00834 Zarfasheen Zia
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Post-Op Complication
Keywords: Abdominal hysterectomy; postoperative pain; Early rehabilitation; Postoperative recovery profile
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative | interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated at the same time following their respective protocols
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Rehab Group (Experimental): The experimental group will receive early physical therapy interventions including patient education, ambulation, in-bed exercises, deep breathing exercises, connective tissue manipulation and TENS during the first 3 post-operative days following abdominal hysterectomy
  Interventions: Other: Advanced early Rehabilitation Program
- Early ambulation Group (Active Comparator): Participants of this group will receive patient education and early ambulation during the first 3 post-operative days following abdominal hysterectomy
  Interventions: Other: Early ambulation

INTERVENTIONS:
Other: Advanced early Rehabilitation Program — Patient education, Ambulation, In bed exercises, Deep breathing exercises: (5 rep x 3set), Connective tissue manipulation for intestinal motility (5 min) and TENS* for incisional pain (30min)
  Arms: Advanced Rehab Group
Other: Early ambulation — Patient education & Assisted ambulation out of bed including walking away from bedside for at least 15 min gradually moving to Unsupervised ambulation for 30 min
  Arms: Early ambulation Group

SUMMARY:
Variety of physical therapy treatments have been used after open abdominal surgery to improve cardiopulmonary and physical function as well as to reduce the incidence of postoperative pulmonary complications. This study intends to determine the effect of early physical therapy interventions on post-operative recovery profile, post-operative ileus and incisional pain following abdominal hysterectomy.

DETAILED DESCRIPTION:
This study is randomized controlled trial which will be conducted at in-patient gynecology department of Pakistan Railway hospital. This study would include total of 42 participants divided into two groups with 21 participants in each group calculated through OpenEpi (CI=95%Power=80%). Individuals will be screened according to inclusion and exclusion criteria and allocated randomly into two groups through sealed envelope method. Experimental group will receive early physical therapy interventions including patient education, ambulation, in-bed exercises, deep breathing exercises, connective tissue manipulation and TENS during the first 3 post-operative days following abdominal hysterectomy. While the control group will receive patient education and early ambulation during the first 3 post-operative days following abdominal hysterectomy.

Post-operative recovery will be assessed on 3rd post-operative day. Intensity of pain will be measured on baseline and 3rd post-operative day. The effect of intervention on post-operative ileus will be measured by monitoring each participant's time to tolerance of oral diet, first passage of stool and flatus

ELIGIBILITY:
Inclusion Criteria:

* open abdominal hysterectomy
* Patient awake and responsive, stable blood pressure, stable heart rate, no dyspnea at rest and pain score < 8 on visual analogue scale on first post-operative day.
* No limitation on physical activities due to any medical problem or restriction by the physician.

Exclusion Criteria:

* Other hysterectomy procedures i.e. laparoscopic or vaginal hysterectomy.
* Females with diabetes or cancer of metastatic nature.
* Neurological or cognitive deficit.
* Ongoing respiratory problem prior to initiation of physical therapy session.
* Medical recommendation not to participate in early active rehabilitation

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients after abdominal hysterectomies will be recruited.
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative recovery profile questionnaire | Post 3rd day
  For hospitalized patients a 17-item version of the PRP will be used (excluding the items "Re-establishing everyday life" and "Sexual activity"). The global score ranges from 0 to 17.
Numeric pain rating scale (NPRS) | Baseline
  Numeric pain rating scale (NPRS) will be used for evaluating intensity of the incisional pain. Its scores range from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric pain rating scale (NPRS) | Post 3rd day
  Numeric pain rating scale (NPRS) will be used for evaluating intensity of the incisional pain. Its scores range from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citak Karakaya I, Yuksel I, Akbayrak T, Demirturk F, Karakaya MG, Ozyuncu O, Beksac S. Effects of physiotherapy on pain and functional activities after cesarean delivery. Arch Gynecol Obstet. 2012 Mar;285(3):621-7. doi: 10.1007/s00404-011-2037-0. Epub 2011 Aug 10. PMID 21830007
- [Background] Allvin R, Svensson E, Rawal N, Ehnfors M, Kling AM, Idvall E. The Postoperative Recovery Profile (PRP) - a multidimensional questionnaire for evaluation of recovery profiles. J Eval Clin Pract. 2011 Apr;17(2):236-43. doi: 10.1111/j.1365-2753.2010.01428.x. Epub 2010 Sep 16. PMID 20846316
- [Background] Mackay MR, Ellis E, Johnston C. Randomised clinical trial of physiotherapy after open abdominal surgery in high risk patients. Aust J Physiother. 2005;51(3):151-9. doi: 10.1016/s0004-9514(05)70021-0. PMID 16137240
- [Background] Hanekom SD, Brooks D, Denehy L, Fagevik-Olsen M, Hardcastle TC, Manie S, Louw Q. Reaching consensus on the physiotherapeutic management of patients following upper abdominal surgery: a pragmatic approach to interpret equivocal evidence. BMC Med Inform Decis Mak. 2012 Feb 6;12:5. doi: 10.1186/1472-6947-12-5. PMID 22309427
- [Background] Reeve JC, Boden I. The physiotherapy management of patients undergoing abdominal surgery. New Zealand Journal of Physiotherapy. 2016;44(1).
- [Background] Castelino T, Fiore JF Jr, Niculiseanu P, Landry T, Augustin B, Feldman LS. The effect of early mobilization protocols on postoperative outcomes following abdominal and thoracic surgery: A systematic review. Surgery. 2016 Apr;159(4):991-1003. doi: 10.1016/j.surg.2015.11.029. Epub 2016 Jan 21. PMID 26804821